CLINICAL TRIAL: NCT02391038
Title: A Phase 1/2 Trial of MLN0264 in Previously Treated Asian Patients With Advanced Gastrointestinal (GI) Carcinoma (Phase 1) or Metastatic or Recurrent Gastric or Gastroesophageal Junction Adenocarcinoma (Phase 2) Expressing Guanylyl Cyclase C (GCC)
Brief Title: MLN0264 in Previously Treated Asian Participants With Advanced Gastrointestinal Carcinoma or Metastatic or Recurrent Gastric or Gastroesophageal Junction Adenocarcinoma Expressing Guanylyl Cyclase C
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated because preliminary PK and overall clinical data demonstrated compelling similarity between Western and Asian participant populations.
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C26004; U1111-1164-1438 (Other: WHO); JapicCTI-152851 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-11-28; First posted 2015-03-18 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Advanced Gastrointestinal Carcinoma; Gastroesophageal Junction Adenocarcinoma; Recurrent Gastric Adenocarcinoma; Recurrent Gastroesophageal Junction Adenocarcinoma; Metastatic Gastric Adenocarcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Recurrent Gastrointestinal Carcinoma
Keywords: MLN0264; Advanced gastrointestinal carcinoma
MeSH Terms: interventions — indusatumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MLN0264 (Experimental): Phase 1: MLN0264 1.2 milligram per kilogram (mg/kg) starting dose, Intravenous (IV), on Day 1 of 3 week cycles, for up to 1 year or until disease progression or unacceptable toxicity. Dosage of MLN0264 will be increased to 1.5 mg/kg then 1.8 mg/kg using a 3 + 3 dose escalation design to determine a maximum tolerated dose (MTD) and/or recommended Phase 2 Dose (RP2D).
  Phase 2: MLN0264, IV, on Day 1 of 3 week cycles, for up to 1 year or until disease progression or unacceptable toxicity. Dosage for this phase will be determined from results of Phase 1 MTD/RP2D.
  Interventions: Drug: MLN0264

INTERVENTIONS:
Drug: MLN0264 — MLN0264 IV.

SUMMARY:
The purpose of this study is to evaluate the effects of MLN0264 in previously treated Asian participants with Advanced Gastrointestinal (GI) Carcinoma (Phase 1) or Metastatic or Recurrent Gastric or Gastroesophageal Junction Adenocarcinoma (Phase 2) Expressing Guanylyl Cyclase C (GCC).

DETAILED DESCRIPTION:
The drug being tested in this study is called MLN0264. This drug is being evaluated to check the effects on previously treated Asian individuals with Advanced GI Carcinoma (Phase 1) or Metastatic or Recurrent Gastric or Gastroesophageal Junction Adenocarcinoma (Phase 2). The study will enroll approximately 95 participants.

In Phase 1, approximately 14 Asian participants with GI malignancies will be enrolled in 3 planned dose cohorts according to the traditional 3 + 3 dose escalation scheme. The starting dose will be 1.2 mg/kg of MLN0264 administered IV on Day 1 of 3-week cycles for up to 1 year or until disease progression or unacceptable toxicity occurs. Dose escalation will take place until Phase 2 recommended dose is determined.

In Phase 2, eligible Asian participants with advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction will be enrolled. Participants must have failed at least 2 lines of prior anticancer therapy for advanced or metastatic disease. Disease recurrence within 6 months of the last dose of post-surgical adjuvant chemotherapy counts as 1 line of prior anticancer therapy for advanced disease.

This multi-center trial will be conducted in Japan, Korea and Taiwan. The overall time to participate in this study is up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Has Diagnosis of GI carcinoma with Immunohistochemistry/ Immunohistochemical (IHC) evidence of expression of GCC protein (H-score of 10 or greater), for which standard treatment is no longer effective or does not offer curative or life-prolonging potential.
* Has completed prior chemotherapy, immunotherapy or radiation therapy at least 4 weeks prior to enrollment (except for Avastin [bevacizumab] for which at least 8 weeks from its last administration should elapse prior to enrollment).
* Histologically confirmed metastatic or advanced inoperable adenocarcinoma of the stomach or gastroesophageal junction with IHC evidence of expression of GCC indicated by an H-score of 10 or greater.
* Has completed prior chemotherapy, immunotherapy or radiation therapy at least 4 weeks prior to enrollment.
* Has measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines.
* Has Eastern Cooperative Oncology Group performance status of 0 or 1 (within 14 days prior to enrollment).
* Females must be 1-year postmenopausal, or even if surgically sterile, agree to use other acceptable forms of birth control.
* Has adequate organ and hematological function.
* Has resolution of all toxic effects of prior treatments except alopecia to Grade 0 or 1 by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03

Exclusion Criteria:

* Has Concurrent treatment or treatment within 4 weeks of study entry with any other investigational agent.
* Female participants who are in the lactation period, even if they discontinue breastfeeding, or have a positive pregnancy test during the Screening period.
* Has uncontrolled, clinically significant, symptomatic cardiovascular disease within 6 months prior to enrollment.
* Has treatment with any medication that has a clinically relevant potential risk of prolonging the QT interval or inducing Torsades de Pointes that cannot be discontinued or switched to a different medication prior to starting study drug.
* Participants with electrocardiogram (ECG) abnormalities considered by the investigator to be clinically -significant, or repeated baseline prolongation of the rate-corrected QT interval millisecond (msec) of electrocardiograph (QTc).
* Ongoing or clinically significant active infection.
* Has signs of peripheral neuropathy.
* Concomitant chemotherapy, hormonal therapy, immunotherapy, or any other form of cancer treatment.
* Use of strong cytochrome P450 (CYP) 3A4 inhibitors within 2 weeks before the first dose of study drug.
* Has any preexisting medical condition of sufficient severity to prevent full compliance with the study.
* Has past or concurrent history of neoplasm other than GI carcinoma (phase 1) or gastric adenocarcinoma (phase 2), except for curatively treated nonmelanoma skin cancer or in situ carcinoma of the cervix uteri.
* Known diagnosis of human immunodeficiency virus (HIV) infection.
* Has asymptomatic brain metastases.
* Has an alcohol or substance abuse disorder.
* Has positive test for hepatitis B surface antigen.
* History of hypersensitivity to any ingredient of MLN0264.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (4):
- Japan (2):
  - Kashiwa-shi, Chiba
  - Minatoku, Tokyo-To
- Seoul, Gyeonggi-do, South Korea
- Taipei, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in Korea, Japan, and Taiwan from 1 December 2014 to 7 October 2015. The study was terminated during the dose-escalation portion of phase 1 and phase 2 was not initiated.
Pre-assignment Details: Participants with a historical diagnosis of gastrointestinal carcinoma were enrolled in 1 of 3 treatment groups: MLN0264 1.2 milligram per kilogram (mg/kg), MLN0264 1.5 mg/kg or MLN0264 1.8 mg/kg during Phase 1.
Groups:
- Phase 1: MLN0264 1.2 mg/kg: MLN0264 1.2 mg/kg, infusion, intravenously over 30 minutes, on Day 1 of every 3 week cycle during the Phase 1, for up to 1 year or until disease progression or unacceptable toxicity
- Phase 1: MLN0264 1.5 mg/kg: MLN0264 1.5 mg/kg, infusion, intravenously over 30 minutes, on Day 1 of every 3 week cycle during the Phase 1, for up to 1 year or until disease progression or unacceptable toxicity
- Phase 1: MLN0264 1.8 mg/kg: MLN0264 1.8 mg/kg, infusion, intravenously, over 30 minutes on Day 1 of every 3 week cycle during the Phase 1, for up to 1 year or until disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Started | 3 | 3 | 6
Completed | 0 | 0 | 0
Not Completed | 3 | 3 | 6
Not completed — Progressive disease | 3 | 3 | 6

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any amount of study drug.
Groups:
- Phase 1: All Participants: Participants who either received MLN0264 1.2 mg/kg as starting dose, or 1.5 mg/kg, or 1.8 mg/kg infusion, intravenously over 30 minutes, on Day 1 of every 3 week cycle of Phase 1, for up to 1 year or until disease progression or unacceptable toxicity.
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 12
Age, Customized [Number; unit: participants]
  Between 45 to 78 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 4
  Taiwan | 1
  Korea, Republic of | 7
Histological classification [Number; unit: participants] — Histological classification included moderately differentiated adenocarcinoma (colon and rectal cancer); intestinal type adenocarcinoma (gastric cancer); adenocarcinoma with lymphovascular invasion; invasive ductal carcinoma of the pancreas, moderately differentiated ductal adenocarcinoma, adenocarcinoma not otherwise specified, tubular adenocarcinoma, and moderately differentiated adenocarcinoma of the transverse and descending colon.
  participants
    Colon cancer | 2
    Rectal cancer | 2
    Gastric cancer | 2
    Lymphovascular invasion | 1
    Invasive ductal carcinoma of the pancreas | 1
    Moderately differentiated ductal adenocarcinoma | 1
    Adenocarcinoma not otherwise specified | 1
    Tubular adenocarcinoma | 1
    Moderately differentiated and descending colon | 1
Participants With Prior Medical Condition [Number; unit: participants] | 12
Participants With Surgical History [Number; unit: participants]
  With Surgical History | 8
  Without Surgical History | 4
Participants With Prior Anticancer Therapy [Number; unit: participants] | 12
Participants With Prior Radiation Therapy [Number; unit: participants]
  With prior radiation therapy | 2
  Without prior radiation therapy | 10
Eastern Cooperative Oncology Group (ECOG) Therapy [Number; unit: participants] — ECOG performance status is used to assess how the disease affects the daily living abilities of the participant. It ranges on the scale from 0-5 (0= normal activity; 1= symptoms but ambulatory; 2= in bed for less than (<) 50 percent (%) of the time; 3= in bed for greater than (>) 50% of the time; 4= 100% bedridden; 5= dead.
  participants
    0 | 8
    1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase 1- Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAE)
Time Frame: Phase 1: Baseline through 30 days after the last dose of study drug (approximately up to 35 weeks)
Population: Safety population includes all participants who received any amount of study drug.
Measure: Number; unit: participants
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 12
participants | 10

2. Primary Outcome: Phase 1- Number of Participants Reporting One or More Serious Adverse Events (SAE)
Time Frame: Phase 1: Baseline through 30 days after the last dose of study drug (Approximately up to 35 weeks)
Population: Safety population included all participants who received any amount of study drug.
Measure: Number; unit: participants
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 12
participants | 4

3. Primary Outcome: Phase 1- Number of Participants Experiencing Dose-limiting Toxicities (DLTs)
Description: Toxicity evaluated as per NationalCancerInstituteCommonTerminologyCriteria for AEs (NCI CTCAE),version 4.03.DLT=any event related to MLN0264:Grade 4 neutropenia(absolute neutrophil count[ANC]less than[<]500 cells/millimeter[mm]^3); >=Grade 3 neutropenia with fever/infection;Grade 4 thrombocytopenia(platelets <25,000/mm^3)/requires platelet transfusion(with/without hemorrhage);Grade 3/greater thrombocytopenia with clinically meaningful bleeding;Anemia requiring blood transfusion;>=Grade 3 nausea/emesis occurring despite using optimal anti-emetic prophylaxis;>=Grade 3 diarrhea despite optimal supportive care measures;any other >=Grade 3 nonhematologic toxicity except brief(<1 week)Grade 3 fatigue;Inability to start next therapy cycle greater than (>)2 weeks due to delayed treatment and adequate recovery of MLN0264-related hematologic or nonhematologic toxicity;other>= Grade 2 MLN0264-related nonhematologic toxicity which requires dose reduction or discontinuation of therapy.
Time Frame: Phase 1: Up to Cycle 1 (3 weeks)
Population: The DLT-Evaluable population included all participants who either experienced DLT during Cycle 1 or received their scheduled Cycle 1 dose and completed all study procedures in Cycle 1 without DLT.
Measure: Number; unit: participants
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 12
participants | 0

4. Primary Outcome: Phase 1- Number of Participants With Markedly Abnormal Laboratory Values
Description: The number of participants with any markedly abnormal standard safety laboratory values collected throughout study. Laboratory assessment includes serum chemistry, hematology, urine analysis and coagulation.
Time Frame: Phase 1: Baseline through 30 days after the last dose of study drug (Approximately up to 35 weeks)
Population: Safety population included all participants who received any amount of study drug.
Measure: Number; unit: participants
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 12
participants
  Serum Chemistry | 10
  Hematology | 12
  Urinalysis | 1
  Coagulation | 5

5. Primary Outcome: Phase 1- Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs include body temperature (oral or tympanic measurement), sitting blood pressure (after the participant has rested for at least 5 minutes), and pulse (beats per minute [bpm]).
Time Frame: Phase 1: Baseline through 30 days after the last dose of study drug (Approximately up to 35 weeks)
Population: Safety population included all participants who received any amount of study drug.
Measure: Number; unit: participants
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 12
participants | 0

6. Primary Outcome: Phase 1- Recommended Phase 2 Dose (RP2D)
Description: RP2D is maximum tolerated dose(MTD) in study Phase1.MTD was highest dose of MLN0264 given at which <=1 of 6 participants experienced DLTduring Cycle1 of Phase1.DLT=any event related to MLN0264:Grade 4 neutropenia ANC less than<500 cells mm^3;>=Grade 3 neutropenia with fever/infection;Grade 4 thrombocytopenia(platelets <25,000/mm^3)/requires platelet transfusion(with/without hemorrhage);Grade 3/greater thrombocytopenia with clinically meaningful bleeding;Anemia requiring blood transfusion;>=Grade 3 nausea/emesis occurring despite using optimal anti-emetic prophylaxis;>=Grade 3 diarrhea despite optimal supportive care measures;any other >=Grade 3 nonhematologic toxicity except brief(<1 week)Grade 3 fatigue;Inability to start next therapy cycle>2 weeks due to delayed treatment and adequate recovery of MLN0264-related hematologic or nonhematologic toxicity;other>= Grade 2 MLN0264-related nonhematologic toxicity which requires dose reduction or discontinuation of therapy.
Time Frame: Phase 1: Baseline through 30 days after the last dose of study drug (Approximately up to 35 weeks)
Population: as for outcome 3
Measure: Number; unit: mg/kg
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 12
mg/kg | NA — None of the participants experienced DLT. Consequently, an evaluation of these participants did not establish RP2D.

7. Primary Outcome: Phase 1: Cycle 1- Cmax: Maximum Observed Plasma Concentration for MLN0264
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: The Pharmacokinetic (PK) evaluable population included all participants who received greater than or equal to (>=1) dose of MLN0264 and had sufficient MLN0264 concentration time data to permit reliable estimation of MLN0264 exposure.
Measure: Geometric Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 6
microgram per milliliter (mcg/mL) | 25.62 (0.907) | 33.84 (6.275) | 35.77 (7.342)

8. Primary Outcome: Phase 1: Cycle 2- Cmax: Maximum Observed Plasma Concentration for MLN0264
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: The PK evaluable population included all participants who received >=1 dose of MLN0264 and had sufficient MLN0264 concentration time data to permit reliable estimation of MLN0264 exposure where Cycle 2 Day 1 PK assessment were available.
Measure: Geometric Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
mcg/mL | 20.99 (0.755) | 29.46 (9.180) | 31.11 (6.874)

9. Primary Outcome: Phase 1: Cycle 1- Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for MLN0264
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: The PK evaluable population included all participants who received >=1 dose of MLN0264 and had sufficient MLN0264 concentration time data to permit reliable estimation of MLN0264 exposure.
Measure: Median (Full Range); unit: day
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 6
day | 0.03 [0.02 to 0.03] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.03]

10. Primary Outcome: Phase 1: Cycle 2- Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for MLN0264
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 8
Measure: Median (Full Range); unit: day
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
day | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.03]

11. Primary Outcome: Phase 1: Cycle 1- AUCinf: Area Under the Concentration-time Curve From Time 0 to Infinity (AUCinf) for MLN0264
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: The PK evaluable population included all participants who received >=1 dose of MLN0264 and had sufficient MLN0264 concentration time data to permit reliable estimation of MLN0264 exposure where Cycle 1 Day 1 PK assessment were available.
Measure: Geometric Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 2 | 3 | 4
day*mcg/mL | 42.97 (4.667) | 63.58 (6.444) | 60.09 (7.330)

12. Primary Outcome: Phase 1: Cycle 2- AUCinf: Area Under the Concentration-time Curve From Time 0 to Infinity (AUCinf) for MLN0264
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 8
Measure: Geometric Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 2 | 1 | 2
day*mcg/mL | 31.81 (11.314) | 74.40 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 61.52 (18.880)

13. Primary Outcome: Phase 1: Cycle 1- AUCint: Area Under the Serum/Plasma Concentration-time Curve From Time 0 to End of the 21-day Dosing Interval (AUCint) for MLN0264
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 2 | 3 | 4
day*mcg/mL | 41.37 (4.667) | 59.63 (6.902) | 57.88 (7.032)

14. Primary Outcome: Phase 1: Cycle 2- AUCint: Area Under the Serum/Plasma Concentration-time Curve From Time 0 to End of the 21-day Dosing Interval (AUCint) for MLN0264
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: The PK evaluable population included all participants who received >=1 dose of MLN0264 and had sufficient MLN0264 concentration time data to permit reliable estimation of MLN0264 exposure where Cycle 2 Day 1 PK assessment were available. Data is not reported for MLN0264 1.2 mg/kg arm as none of the participants had data evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 0 | 1 | 2
day*mcg/mL |  | 71.60 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 58.03 (19.233)

15. Primary Outcome: Phase 1: Cycle 1- Ctrough: Observed Concentration Measured at the End of a Dosing Interval for MLN0264
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 2 | 3 | 4
mcg/mL | 0.201 (0.0113) | 0.309 (0.0490) | 0.261 (0.0831)

16. Primary Outcome: Phase 1: Cycle 2- Ctrough: Observed Concentration Measured at the End of a Dosing Interval for MLN0264
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 0 | 1 | 2
mcg/mL |  | 0.365 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 0.369 (0.0283)

17. Primary Outcome: Phase 1: Cycle 1- Cmax: Maximum Observed Serum Concentration for Total Antibody (TAb)
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: The PK evaluable population included all participants who received >=1 dose of MLN0264 and had sufficient TAb concentration time data to permit reliable estimation of the PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 6
mcg/mL | 24.53 (2.179) | 32.12 (9.180) | 36.31 (7.709)

18. Primary Outcome: Phase 1: Cycle 2- Cmax: Maximum Observed Serum Concentration for TAb
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: The PK evaluable population included all participants who received >=1 dose of MLN0264 and had sufficient TAb concentration time data to permit reliable estimation of the PK parameters where Cycle 2 Day 1 PK assessment were available.
Measure: Geometric Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
mcg/mL | 24.28 (3.592) | 33.33 (9.454) | 36.54 (6.471)

19. Primary Outcome: Phase 1: Cycle 1- Tmax: Time to Reach the Maximum Serum Concentration (Cmax) for TAb
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 17
Measure: Median (Full Range); unit: day
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 6
day | 0.03 [0.02 to 0.03] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.03]

20. Primary Outcome: Phase 1: Cycle 2- Tmax: Time to Reach the Maximum Serum Concentration (Cmax) for TAb
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 18
Measure: Median (Full Range); unit: day
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
day | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.03]

21. Primary Outcome: Phase 1: Cycle 1- AUCinf: Area Under the Concentration-time Curve From Time 0 to Infinity (AUCinf) for TAb
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: The PK evaluable population included all participants who received >=1 dose of MLN0264 and had sufficient TAb concentration time data to permit reliable estimation of the PK parameters where Cycle 1 Day 1 PK assessment were available.
Measure: Geometric Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 2 | 2 | 3
day*mcg/mL | 68.82 (22.910) | 154.95 (5.657) | 149.65 (31.321)

22. Primary Outcome: Phase 1: Cycle 2- AUCinf: Area Under the Concentration-time Curve From Time 0 to Infinity (AUCinf) for TAb
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: The PK evaluable population included all participants who received >=1 dose of MLN0264 and had sufficient TAb concentration time data to permit reliable estimation of the PK parameters where Cycle 2 Day1 PK assessment were available. Data is not reported for MLN0264 1.2 mg/kg arm because none of the participants had data evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 0 | 1 | 1
day*mcg/mL |  | 192.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 204.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.

23. Primary Outcome: Phase 1: Cycle 1- AUCint: Area Under the Serum/Plasma Concentration-time Curve From Time 0 to End of the 21-day Dosing Interval (AUCint) for TAb
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 21
Measure: Geometric Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
day*mcg/mL | 69.82 (20.647) | 116.59 (20.775) | 112.46 (30.653)

24. Primary Outcome: Phase 1: Cycle 2- AUCint: Area Under the Serum/Plasma Concentration-time Curve From Time 0 to End of the 21-day Dosing Interval (AUCint) for TAb
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 22
Measure: Geometric Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 0 | 1 | 2
day*mcg/mL |  | 164.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 147.21 (32.527)

25. Primary Outcome: Phase 1: Cycle 1- Ctrough: Observed Concentration Measured at the End of a Dosing Interval for TAb
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: The PK evaluable population included all participants who received >=1 dose of MLN0264 and had sufficient TAb concentration time data to permit reliable estimation of the PK parameters where Cycle 1 Day1 PK assessment were available. Data is not reported for MLN0264 1.2 mg/kg arm because none of the participants had data evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
mcg/mL | 0.835 (0.4912) | 1.479 (0.0794) | 1.140 (0.9592)

26. Primary Outcome: Phase 1: Cycle 2- Ctrough: Observed Concentration Measured at the End of a Dosing Interval for TAb
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 22
Measure: Geometric Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 0 | 1 | 2
mcg/mL |  | 2.300 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 2.560 (0.0424)

27. Primary Outcome: Phase 1: Cycle 1- Cmax: Maximum Observed Plasma Concentration for Monomethyl Auristatin E (MMAE)
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: The PK evaluable population included all participants who received >=1 dose of MLN0264 and had sufficient MMAE concentration time data to permit reliable estimation of the PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 6
nanogram per milliliter (ng/mL) | 2.002 (2.9479) | 2.335 (0.3889) | 6.614 (4.6853)

28. Primary Outcome: Phase 1: Cycle 2- Cmax: Maximum Observed Plasma Concentration for MMAE
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: The PK evaluable population included all participants who received >=1 dose of MLN0264 and had sufficient MMAE concentration time data to permit reliable estimation of the PK parameters where Cycle 2 Day 1 PK assessment were available.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
ng/mL | 2.777 (5.0507) | 2.611 (1.1907) | 6.976 (5.6196)

29. Primary Outcome: Phase 1: Cycle 1- Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for MMAE
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 27
Measure: Median (Full Range); unit: day
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 6
day | 2.04 [0.42 to 3.00] | 2.88 [2.84 to 3.00] | 2.45 [1.90 to 3.00]

30. Primary Outcome: Phase 1: Cycle 2- Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for MMAE
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 28
Measure: Median (Full Range); unit: day
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
day | 2.03 [1.90 to 3.00] | 2.00 [2.00 to 2.92] | 2.89 [1.96 to 3.00]

31. Primary Outcome: Phase 1: Cycle 1- AUCinf: Area Under the Concentration-time Curve From Time 0 to Infinity (AUCinf) for MMAE
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: The PK evaluable population included all participants who received >=1 dose of MLN0264 and had sufficient MMAE concentration time data to permit reliable estimation of the PK parameters where Cycle 1 Day 1 PK assessment were available.
Measure: Geometric Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 2 | 3 | 5
day*ng/mL | 8.510 (0.0424) | 17.170 (5.0302) | 53.172 (53.8275)

32. Primary Outcome: Phase 1: Cycle 2- AUCinf: Area Under the Concentration-time Curve From Time 0 to Infinity (AUCinf) for MMAE
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: The PK evaluable population included all participants who received >=1 dose of MLN0264 and had sufficient MMAE concentration time data to permit reliable estimation of the PK parameters where Cycle2 Day1 PK assessment were available. Data is not reported for MLN0264 1.2 mg/kg arm because none of the participants had data evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 0 | 1 | 2
day*ng/mL |  | 16.600 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 37.212 (12.5158)

33. Primary Outcome: Phase 1: Cycle 1- AUCint: Area Under the Serum/Plasma Concentration-time Curve From Time 0 to End of the 21-day Dosing Interval (AUCint) for MMAE
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 31
Measure: Geometric Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
day*ng/mL | 15.846 (27.9611) | 16.840 (4.7596) | 52.327 (51.8349)

34. Primary Outcome: Phase 1: Cycle 2- AUCint: Area Under the Serum/Plasma Concentration-time Curve From Time 0 to End of the 21-day Dosing Interval (AUCint) for MMAE
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 32
Measure: Geometric Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 0 | 1 | 2
day*ng/mL |  | 16.400 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 36.603 (12.1622)

35. Primary Outcome: Phase 1: Cycle 1- Ctrough: Observed Concentration Measured at the End of a Dosing Interval for MMAE
Time Frame: Day 1 of Cycle 1: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 31
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
ng/mL | 0.049 (0.0665) | 0.037 (0.0025) | 0.157 (0.3717)

36. Primary Outcome: Phase 1: Cycle 2- Ctrough: Observed Concentration Measured at the End of a Dosing Interval for MMAE
Time Frame: Day 1 of Cycle 2: predose and at multiple time points (up to 336 hours) post-dose
Population: as for outcome 32
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1: MLN0264 1.2 mg/kg | Phase 1: MLN0264 1.5 mg/kg | Phase 1: MLN0264 1.8 mg/kg
Number analyzed (Participants) | 0 | 1 | 2
ng/mL |  | 0.057 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 0.117 (0.0824)

37. Primary Outcome: Phase 2- Overall Response Rate
Description: ORR is the percentage of participants with complete response [CR] + partial response [PR]) based on modified Response Evaluation Criteria in Solid Tumors (RECIST). Overall response rate (CR + PR) based on modified RECIST version 1.1 guidelines. CR: Disappearance of all target lesions and PR: at least a 30 percentage (%) decrease in the sum of the longest diameter (LD) of target lesions, taking the baseline sum LD as reference. All measurable lesions up to a maximum of 2 lesions per organ, 5 lesions in total representative of all involved organs were identified as target lesions at baseline. Target lesions were selected on the basis of size (longest lesions) and suitability for reproducible repeated measurements.
Time Frame: Baseline until end of study treatment (approximately 1 year)
Population: Data was not reported for this measure as Phase 2 was not initiated, due to study termination during the dose-escalation portion of phase 1 consistent with the findings that preliminary PK and overall clinical data demonstrated compelling similarity between Western and Asian participant populations.
Groups:
- Phase 2: All Participants: MLN0264, infusion was planned to be administered intravenously on Day 1 of every 3 week cycle for up to 1 year or until disease progression or unacceptable toxicity during Phase 2. Dosage for this phase was to be determined from results of Phase 1 MTD/RP2D.
Arm/Group | Phase 2: All Participants
Number analyzed (Participants) | 0

38. Secondary Outcome: Phase 1- Number of Participants With Antitherapeutic Antibodies (ATAs)
Description: Blood samples was collected predose to evaluate ATA. Data was collected only for limited period due to early termination of the study.
Time Frame: Day 1 of Cycle 1, 2, 3, 4: predose
Population: Safety population included all participants who received any amount of study drug.
Measure: Number; unit: participants
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 12
participants | 0

39. Secondary Outcome: Phase 1- Disease Response Based on the Investigator's Assessment
Description: Disease response was based on the investigator's assessment using the modified RECIST version 1.1 guidelines. Evaluation of target lesions included CR (Disappearance of all target lesions),PR(at least a 30% decrease in the sum of the LD of target lesions),Progressive disease (PD:at least a 20% increase in the sum of the LD of target lesions, taking the smallest sum LD recorded as reference since the treatment started or the appearance of one or more new lesions) and Stable disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD).Evaluation of Non target Lesions included CR (disappearance of all non target lesions and normalization of tumor marker level), Incomplete response/SD (Persistence of 1 or more non target lesions and/or maintenance of tumor marker level above the normal limits) and PD(Appearance of 1 or more new lesions and/or unequivocal progression of existing non target lesions).
Time Frame: Phase 1: Day 21 of every other cycle (Cycle 2, 4, 6, 8) up to End of treatment (EOT) (Cycle10 or week 30)
Population: The Response-Evaluable population is defined as all participants with measurable disease who receive at least 1 dose of MLN0264 and have at least 1 post baseline response assessment.
Measure: Number; unit: participants
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 12
participants
  CR | 0
  PR | 0
  SD | 0
  PD | 12

40. Secondary Outcome: Phase 2- Percentage of Participants Who Experience at Least One TEAE
Time Frame: Phase 2: Baseline up to 30 days after last dose of study drug (approximately 1 year)
Population: as for outcome 37
Arm/Group | Phase 2: All Participants
Number analyzed (Participants) | 0

41. Secondary Outcome: Phase 2- Percentage of Participants Who Experience at Least One SAE
Time Frame: Phase 2: Baseline up to 30 days after last dose of study drug (approximately 1 year)
Population: as for outcome 37
Arm/Group | Phase 2: All Participants
Number analyzed (Participants) | 0

42. Secondary Outcome: Phase 2- Number of Participants With Markedly Abnormal Laboratory Values
Description: as for outcome 4
Time Frame: Phase 2: Baseline up to 30 days after last dose of study drug (approximately 1 year)
Population: as for outcome 37
Arm/Group | Phase 2: All Participants
Number analyzed (Participants) | 0

43. Secondary Outcome: Phase 2- Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: as for outcome 5
Time Frame: Phase 2: Baseline up to 30 days after last dose of study drug (approximately 1 year)
Population: as for outcome 37
Arm/Group | Phase 2: All Participants
Number analyzed (Participants) | 0

44. Secondary Outcome: Phase 2- Progression-free Survival (PFS)
Description: PFS is defined as the time from the date of first study drug administration to the date of first documentation of progressive disease or death. For a participant who has not progressed and is last known to be alive, PFS was censored at the last response assessment that was stable disease or better. PD:at least a 20% increase in the sum of the LD of target lesions, taking the smallest sum LD recorded as reference since the treatment started or the appearance of one or more new lesions.
Time Frame: Baseline up to EOT, thereafter every 12 weeks until the occurrence of PD, the start of subsequent antineoplastic therapy, or 6 months after discontinuation from treatment, whichever occurs first (total duration of assessment up to 1.5 years)
Population: as for outcome 37
Arm/Group | Phase 2: All Participants
Number analyzed (Participants) | 0

45. Secondary Outcome: Phase 2- Duration of Response (DOR)
Description: DOR is defined as the time from the date of first documentation of a confirmed response to the date of first documentation of Progressive Disease (PD). Responders without documentation of PD were censored at the last response assessment that was stable disease or better. CR: disappearance of all target lesions; PR: at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD and PD:at least a 20% increase in the sum of the LD of target lesions, taking the smallest sum LD recorded as reference since the treatment started or the appearance of one or more new lesions.
Time Frame: Day 21 of every other cycle (Cycle 2, 4, 6, 8) up to EOT (approximately 1 year)
Population: as for outcome 37
Arm/Group | Phase 2: All Participants
Number analyzed (Participants) | 0

46. Secondary Outcome: Phase 2- Disease Control Rate (DCR)
Description: DCR is defined as Complete Response (CR) rate + Partial Response (PR) rate + stable disease (SD) rate with a minimum of 12 weeks' duration. Duration of SD is defined as the time from the date of first study drug administration to the date of first documentation of disease progression for participants who achieved SD as the best overall response. CR: disappearance of all target lesions; PR: at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; PD:at least a 20% increase in the sum of the LD of target lesions, taking the smallest sum LD recorded as reference since the treatment started or the appearance of one or more new lesions) and SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Phase 2: Day 21 of every other cycle (Cycle 2, 4, 6, 8) up to EOT (approximately 1 year)
Population: as for outcome 37
Arm/Group | Phase 2: All Participants
Number analyzed (Participants) | 0

47. Secondary Outcome: Phase 2- Overall Survival (OS)
Description: OS is defined as the time from the date of first study drug administration to the date of death. Participants without documentation of death at the time of analysis were censored at the date when they were last known to be alive.
Time Frame: Baseline up to EOT thereafter every 12 weeks until death or the start of subsequent antineoplastic therapy, or 6 months after discontinuation from treatment, whichever occurs first (total duration of assessment up to 1.5 years)
Population: as for outcome 37
Arm/Group | Phase 2: All Participants
Number analyzed (Participants) | 0

48. Secondary Outcome: Phase 2- Plasma Concentration of MLN0264
Time Frame: Day 1 of every cycle (up to 1 year): predose and at multiple time points(up to 336 hours) post-dose
Population: as for outcome 37
Arm/Group | Phase 2: All Participants
Number analyzed (Participants) | 0

49. Secondary Outcome: Phase 2- Tumor Size Reduction
Description: For each participant, the best percentage of tumor reduction from baseline in the sum of the diameter was calculated.
Time Frame: Baseline up to approximately 1 year
Population: as for outcome 37
Arm/Group | Phase 2: All Participants
Number analyzed (Participants) | 0

50. Secondary Outcome: Phase 2- Guanylyl Cyclase C (GCC) H-score Assessed by Immunohistochemistry (IHC)
Description: The H-score is a method of assessing the extent of nuclear immunoreactivity, applicable to steroid receptors. The score is obtained by the formula: 3 * percentage of strongly staining nuclei + 2 * percentage of moderately staining nuclei + percentage of weakly staining nuclei, giving a range of 0 to 300. The 600 H-score is based on the sum of the 0 to 300 H-score for cytoplasmic staining and the 0 to 300 H-score for apical staining
Time Frame: Baseline up to approximately 1 year
Population: as for outcome 37
Groups:
- Phase 2: All Participants: MLN0264, injection, intravenously on Day 1 of 3 week cycles of Phase 2, until disease progression or unacceptable toxicity. Dosage for this phase was determined from results of Phase 1 MTD/RP2D.
Arm/Group | Phase 2: All Participants
Number analyzed (Participants) | 0

51. Secondary Outcome: Phase 2- Number of Participants With ATA in Serum
Description: Blood samples were to be collected predose to evaluate ATA.
Time Frame: Baseline up to approximately 1 year
Population: as for outcome 37
Arm/Group | Phase 2: All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug through 30 days after the last dose of any study drug (approximately 35 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Phase 1: All Participants
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: All Participants (N=12)
Tumor hemorrhage and ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Asthenia (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: All Participants (N=12)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Eye discharge (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 2
Fatigue (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 2
Herpes zoster (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.